CLINICAL TRIAL: NCT00539734
Title: Electrophysiologic Changes After Intravitreal Ranibizumab (Lucentis) for Age-related Macular Degeneration
Brief Title: Changes in Retinal Function After Intravitreal Ranibizumab for Age-related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Dr.Patama Bhurayanontachai, Prince of Songkla University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50/362-003-2
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2011-04-08 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Age-related Macular Degeneration
Keywords: age-related macular degeneration (AMD); choroidal neovascularization membrane(CNVM); ranibizumab; anti-vascular endothelial growth factor; electrophysiology; electroretinography
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ranibizumab — A single dose of 0.5 mg ranibizumab injected intravitreally.
  Other Names: Lucentis

SUMMARY:
Age-related macular degeneration, a leading cause of blindness, is caused by an abnormal growth of the vessels beneath the retina. Ranibizumab (Lucentis) is a new drug that inhibits the growth of new vessels and has recently been approved by FDA for treating this condition. This study is carried out to evaluate the changes in retinal function after an injection of ranibizumab.

DETAILED DESCRIPTION:
The functional changes of the retina can be recorded by an electroretinography (ERG).

ELIGIBILITY:
Inclusion Criteria:

* Age 45 years and above
* Clinical diagnosis of wet AMD
* First injection of ranibizumab protocol
* Best corrected visual acuity 20/32 - 20/320
* Consent form obtained

Exclusion Criteria:

* Previously treated wet AMD patients
* Patients with other ocular diseases which can cause abnormal ERG such as glaucoma, uveitis or retinitis pigmentosa, etc.
* Pregnancy
* History of seizure

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patama Bhurayanontachai, MD, Principal Investigator — Department of Ophthalmology, Faculty of Medicine, Prince of Songkla University
Locations (1):
- Department of Ophthalmology, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Kaiser PK, Brown DM, Zhang K, Hudson HL, Holz FG, Shapiro H, Schneider S, Acharya NR. Ranibizumab for predominantly classic neovascular age-related macular degeneration: subgroup analysis of first-year ANCHOR results. Am J Ophthalmol. 2007 Dec;144(6):850-857. doi: 10.1016/j.ajo.2007.08.012. Epub 2007 Oct 22. PMID 17949673

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab Group: Ranibizumab 0.5 mg (Lucentis®; Novartis Pharma AG, Basel, Switzerland) was injected intravitreally at 4.0 mm from the limbus in phakic eyes and at 3.5 mm in pseudophakic eyes. Re-treatment with the interval of a month apart is considered under the retinal condition.
Period: Overall Study
Arm/Group | Ranibizumab Group
Started | 26
Completed | 25
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ranibizumab Group
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 66.5 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 10
Region of Enrollment [Number; unit: participants]
  Thailand | 26

OUTCOME MEASURES:

1. Primary Outcome: Height (Amplitude) of Multifocal ERG Signal
Description: Comparing the response in hight of signal amplitude at 3 months after treatment with baseline data.
Time Frame: baseline, 3 months
Population: Analysis was per protocol
Measure: Mean (Standard Deviation); unit: nanovolt/degree^2
Units Other Than Participants: eyes
Arm/Group | Ranibizumab Group
Number analyzed (Participants) | 25
Number analyzed (eyes) | 26
nanovolt/degree^2 | 2.859 (1.085)
Statistical Analysis 1: Comparison: Ranibizumab Group; Comparing pre-operative data with postoperative data in terms of changes in amplitude height and implicit time; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Postoperative Complication
Description: For instance, Endophthalmitis, retinal detachment
Time Frame: 1 month
Reporting Status: Not Posted

3. Primary Outcome: Time to Response (Implicit Time) of Multifocal ERG Signal
Description: Comparing the change in time of signal response (implicit time) at 3 months after treatment with baseline data.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: millisecond
Units Other Than Participants: eyes
Arm/Group | Ranibizumab Group
Number analyzed (Participants) | 25
Number analyzed (eyes) | 26
millisecond | 31.621 (3.563)

ADVERSE EVENTS:
Arm/Group | Ranibizumab Group
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

LIMITATIONS AND CAVEATS:
Small number of participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes